CLINICAL TRIAL: NCT02774200
Title: A One-arm Exploratory Clinical Research Program Study of Apatinib in Advanced Metastatic Renal Cell Carcinoma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HBR001
Record Dates: First submitted 2016-05-11; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-03

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- test group (Experimental): Apatinib 500 mg, po, qd, continuous medication for a period of eight weeks.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib 500 mg, po, qd, continuous medication for a period of eight weeks.
  Other Names: Apatinib Mesylate Tablets

SUMMARY:
A one-arm exploratory clinical research program Study of Apatinib in Advanced Metastatic Renal Cell Carcinoma （mRCC） Patients.It's arm to evaluate the treatment of advanced metastatic renal cell carcinoma in patients with objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), overall survival (OS), quality of life score (QoL) and safety.

DETAILED DESCRIPTION:
Objective response rate (ORR), disease control rate (DCR) (according to RECIST 1.1 Standard Edition)，progression-free survival (PFS), overall survival (OS), quality of life (QoL).Evaluation once every 8 weeks, If the efficacy results of the evaluation are complete response (CR) or partial response (PR), confirmed imaging efficacy at 4 weeks after the initial assessment ， efficacy evaluation time window of ± 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to 75 years
* Histologically or cytologically confirmation with a renal clear cell histologic component and metastases
* Presence of a single diameter measurable lesions (eg, ≥1 malignant tumors with at least one single diameter can be accurately measured, conventional computer tomography scan [CT] or magnetic resonance [MRI] requires at least one path ≥20mm, if the interphase reconstruction of spiral computed tomography scan ≤5mm [CT], at least one path ≥10mm). Bone lesions, ascites, peritoneal metastasis or miliary lesions, pleural or pericardial effusion, skin or lung lymphangitis, cystic lesion or lesions after radiotherapy is not measurable lesion
* Life expectancy more than 3 months
* The progress of the disease must be according to RECIST criteria (version 1.0) after a previous systemic treatment of first-line metastatic renal cell carcinoma. Previous treatment program includes one or more of the following drugs: Sunitinib, Sorafenib, Bevacizumab + Interferon-α (IFN-α), Temsirolimus or Cytokine;
* Adequate organ function, defined as follows: the absolute number of Neutrophil (ANC) same or more than 1500 cells / mm3; Platelet same or more than 75,000 cells / mm3; Hemoglobin same or more than 9.0 g / dL; Aspartate aminotransferase（AST）and alanine aminotransferase (ALT) same or less than equal 2.5 x upper limit normal (xULN), if liver metastases, Aspartate aminotransferase (AST) and ALT same or less than 5.0 times ULN;Total bilirubin same or less than 1.5 times ULN，Serum Creatinine same or less than 1.5 times ULN, Creatinine clearance same or more than 60 mL/min, Urinary dipstick proteinuria <2+. If the urine protein same or more than 2+, the need for 24-hour urinary protein excretion, and 24-hour urine protein <2 g
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* The prior systemic therapy, radiation therapy, surgery at least two weeks apart (bevacizumab + IFN-α therapy for at least 4 weeks apart), all treatment-related toxicity recovered to ≤1 grade defined according to 3.0 versions of NCI CTCAE defined, or recovered to baseline levels, except for alopecia, or hypothyroidism
* The measured value of twice baseline blood pressure (interval of at least 1 hour) show inexistent Hypertension that cannot be controlled by medication. Baseline systolic blood pressure should be same or less than 140 mm Hg, baseline diastolic blood pressure should be same or less than 90 mm Hg. Patients with antihypertensive drugs can be controlled by the group
* For the fertility of women ,the serum or urine pregnancy test must be negative within pre-treatment three days
* Signed and dated informed consent of document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment
* Patient consent and well compliance, scheduled to accept the visits, treatment, laboratory tests and other study procedures

Exclusion Criteria:

* Patients who received more than one first-line for the Metastatic Renal Cell Carcinoma (mRCC) systemic treatment
* Patients who received any neoadjuvant or adjuvant systemic treatment
* Begin to study 4 weeks later than major surgery treatment time, or 2 weeks later than radiotherapy. Allow received palliative radiotherapy for metastatic lesion, but at least one measurable lesions did not receive radiation therapy
* The gastrointestinal tract anomalies

  * unable to take oral medication
  * require intravenous nutrition
  * previous surgical treatment influence drug absorption include total gastrectomy
  * In the past six months have been treated for active ulcer disease
  * In the past three months with cancer unrelated activities gastrointestinal bleeding, including vomiting blood, blood in the stool or black stools, endoscopy or colonoscopy colon without evidence of remission
  * malabsorption syndrome.
* Currently accepted or may need to accept treatment with potent CYP3A4 inhibitors (eg, grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, blessing Secretary amprenavir and delavirdine)
* Currently accepted or may need to accept CYP3A4 or CYP1A2 inducer treatment (eg, carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine , primidone, rifabutin, rifampicin, Hypericum perforatum)
* Need to accept the oral vitamin K antagonists of anticoagulant therapy. Allows the use of low dose of anticoagulant drugs to remain central venous channel unobstructed and prevention of deep vein thrombosis. Allow treatment dose low molecular heparin
* Active epilepsy or brain metastases, spinal cord compression or meningitis carcinomatosa
* Patients who have unable to control the disease or active infection
* Situation appeared within 12 months before with the study drug: myocardial infarction, uncontrolled angina, coronary artery/peripheral artery bypass grafting, with symptoms of congestive heart failure, cerebrovascular accident, transient ischemic attack, deep vein thrombosis or pulmonary embolism within 6 months
* Known history of Human Immunodeficiency Virus(HIV) positive or Immune Deficiency Syndrome(AIDS) related diseases
* Medical History:Have other malignant tumors (except renal cell carcinoma), not including treatable form of skin cancer (non malignant melanoma), breast carcinoma in situ or cervical carcinoma in situ, or any other tumors has been cured, and no evidence of disease recurrence within 2 years
* Patients who are dementia or obvious mental retardation
* Women with pregnancy or lactation, or fertility but during treatment and 6 months after treatment of termination unwilling or unable to use effective contraception to avoid pregnancy patients with male or female
* With other serious acute and chronic physical or mental illness or abnormal laboratory tests, according to the judgment may increase the risk of to participate in research or related to drug treatment, or may affect the interpretation of the results, or other situations that the researchers considered unsuitable for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 8 weeks

SECONDARY OUTCOMES:
progression-free survival (PFS) | 8 weeks
overall survival (OS) | 8 weeks
quality of life score (QoL) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: peng chen, M.D., Principal Investigator — Department of Pulmonary Medical Oncology, Tianjin Medical University Cancer Hospital

IPD SHARING:
Plan to Share IPD: No